CLINICAL TRIAL: NCT04895150
Title: Investigation of Upper Extremity Exercise Capacity, Muscle Oxygenation, Balance and Physical Activity Levels in Patients With Primary Ciliary Dyskinesia
Brief Title: Upper Extremity Exercise Capacity, Muscle Oxygenation, Balance in Patients With Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 408
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Primary Ciliary Dyskinesia; Upper Extremity Exercise Capacity; Muscle Oxygenation; Balance; Physical Activity
MeSH Terms: conditions — Ciliary Motility Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Upper extremity exercise capacity (6 minutes Pegboard and Ring Test), muscle oxygenation ("Moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), balance("Biodex Balance System®" and Y balance test), physical activity level (multi-sensor activity monitor) and quality of life (Quality of Life scale for Primary Ciliary Dyskinesia (QOL-PCD scale version 4.3)) will be evaluated.
- Healthy controls;: Upper extremity exercise capacity (6 minutes Pegboard and Ring Test), muscle oxygenation ("Moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), balance("Biodex Balance System®" and Y balance test), physical activity level (multi-sensor activity monitor) and quality of life (Quality of Life scale for Primary Ciliary Dyskinesia (QOL-PCD scale version 4.3)) will be evaluated.

SUMMARY:
The main aim of the study is to evaluate upper extremity exercise capacity and muscle oxygenation in patients with primary ciliary dyskinesia. The secondary aim of the study is to evaluate respiratory function, respiratory muscle strength and endurance, peripheral muscle strength, balance, physical activity level and quality of life in patients with primary ciliary dyskinesia and compare all parameters with healthy controls.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is a genetic, heterogeneous disease caused by cilia absence or dysfunction. Impaired function of motile cilia leads to impaired mucociliary clearance, recurrent chest infections, and progressive destruction of the lung structure. Clinical features include neonatal respiratory distress syndrome, chronic daily productive cough, chronic nasal congestion, and chronic or recurrent otitis media.

Pulmonary functions, exercise capacity, respiratory muscle strength and endurance, peripheral muscle strength, physical activity level and quality of life were affected in patients. The number of studies on these subjects is limited.

Pulmonary function and extremity muscle strength are determinants of exercise capacity in chronic obstructive pulmonary disease. Decreased strength and endurance in the limb muscles is associated with exercise intolerance. Patients have decreased upper extremity muscle strength. There is no study in the literature evaluating upper extremity exercise capacity in patients with PCD. Measuring the oxygen saturation of cardiorespiratory and peripheral muscles is important for understanding the dynamics of oxygen delivery and consumption during exercise. There are no studies in the literature evaluating muscle oxygenation in this patient population.

The main aim of the study is to evaluate upper extremity exercise capacity and muscle oxygenation in patients with primary ciliary dyskinesia. The secondary aim of the study is to evaluate respiratory function, respiratory muscle strength and endurance, peripheral muscle strength, balance, physical activity level and quality of life in patients with primary ciliary dyskinesia and compare them with healthy controls.

The study was planned cross-sectional. Patients with primary ciliary dyskinesia referred to the Cardiopulmonary Rehabilitation Unit of Gazi University Physiotherapy and Rehabilitation Department by the physicians of the Department of Pediatric Pulmonary Diseases of Gazi University Faculty of Medicine will be included in the study. At least 18 patients with primary ciliary dyskinesia and at least 18 healthy controls of similar age and sex will be evaluated in the study. The assessments will be completed in two days.

Upper extremity exercise capacity (6 minutes Pegboard and Ring Test), muscle oxygenation ("Moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), balance("Biodex Balance System®" and Y balance test), physical activity level (multi-sensor activity monitor) and quality of life (Quality of Life scale for Primary Ciliary Dyskinesia (QOL-PCD scale version 4.3) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* 6-18 years old
* Diagnosed with primary ciliary dyskinesia
* Stability of clinical condition

Healthy controls;

* 6-18 years old

Exclusion Criteria:

Patients;

* Diagnosed neurological, cognitive problem that can affect evaluations,
* Acute pneumonia or any infection
* History of exacerbation in the last 1 month
* More than 10% change in FEV1 in the last 6 months
* History of coronavirus disease (COVID-19)
* History of smoking
* Diagnosed vision, hearing, vestibular, or neurological problems that can affect balance
* Diagnosed orthopedic problems affecting mobility or a history of musculoskeletal surgery

Healthy controls;

* Diagnosed neurological, cognitive problem that can affect evaluations
* Diagnosed vision, hearing, vestibular, or neurological problems that can affect balance
* History of coronavirus disease (COVID-19)
* History of smoking
* Trouble understanding and following the exercise test instruction

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At least 18 patients with primary ciliary dyskinesia will be included in patients group and 18 healthy individuals will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | First Day
  Upper extremity exercise capacity will be evaluated with the six-minute pegboard and ring test (6-PBRT). A pegboard with two upper and lower bars set at participants shoulder level and above the shoulder level will used. Ten rings will placed on both the lower bars. Patients will be asked to move a single ring at a time with both hands from the lower bars to the upper. The score is the total number of rings moved the six-minute period.
Muscle Oxygenation | First Day
  Muscle oxygenation assessment will be performed using the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device will be placed on the 1/3 lower motor point of the quadriceps muscle group of the dominant leg and on the dominant arm deltoid muscle. A minimum of 3 minutes will be waited until the resting measurements and skeletal muscle oxygenation (StO2) signal stabilize. The measurements will be repeated during six minute walking test and six minute pegboard and ring test.

SECONDARY OUTCOMES:
Functional exercise capacity | First Day
  Functional exercise capacity will be evaluated with 6-minute walking test according to the American Thoracic Society and European Respiratory Society criteria.
Balance | Second day
  Static balance assessment will be evaluated using the "Biodex Balance System®". The test period will be 20 seconds, and there will be a 10-second break between evaluations. General stability index, anterior / posterior (AP) stability index, medial / lateral (ML) stability index and their standard deviations will be obtained from the system as a result of the test. The tests will first be carried out on the hard ground with open eyes. The tests will second be carried out on the hard ground with closed eyes. The tests will third be carried out on the soft ground with open eyes. Dynamic balance will be evaluated with the Y balance test.
Physical activity (Total energy expenditure) | Second day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day) | Second day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Respiratory muscle strength | First day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be measured with a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria.
Respiratory muscle endurance | Second Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load. The test will be started with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80% and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period will be recorded.The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced vital capacity (FVC) will be measured.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. FEV1 / FVC will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Peak flow rate (PEF) will be measured.
Life quality | Second day
  Quality of life will be evaluated with the Quality of Life scale for Primary Ciliary Dyskinesia (QOL-PCD scale version 4.3)(Turkish version). The scale have well-established reliability and validity. There are four separate versions of QOL-PCD for three separate age-appropriate.The scale includes questions about physical function, emotional function, social function, respiratory symptoms, treatment burden, hearing symptoms, role, health perceptions, vitality, eating and weight. The scale included sub-groups involving different situations according to the different ages. The total numbers of items in the scale are 37 in the questionnaire for children, 43 in the one for adolescents, 49 in the one for adults, 41 in the parents of the patients in the age group of 6-12 years. Items are rated according to a 4-point scale. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, Prof.Dr., Study Director — Gazi University; Şeyma Mutlu, Pt., Study Chair — Gazi University; Tuğba ŞİŞMANLAR EYÜBOĞLU, Asc.Prof.Dr., Principal Investigator — Gazi University; Ayşe Tana ARSLAN, Prof.Dr., Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Faculty of Health Science, Ankara
  - Gazi University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valerio G, Giallauria F, Montella S, Vaino N, Vigorito C, Mirra V, Santamaria F. Cardiopulmonary assessment in primary ciliary dyskinesia. Eur J Clin Invest. 2012 Jun;42(6):617-22. doi: 10.1111/j.1365-2362.2011.02626.x. Epub 2011 Nov 29. PMID 22121832
- [Background] Ring AM, Buchvald FF, Holgersen MG, Green K, Nielsen KG. Fitness and lung function in children with primary ciliary dyskinesia and cystic fibrosis. Respir Med. 2018 Jun;139:79-85. doi: 10.1016/j.rmed.2018.05.001. Epub 2018 May 3. PMID 29858006
- [Background] Madsen A, Green K, Buchvald F, Hanel B, Nielsen KG. Aerobic fitness in children and young adults with primary ciliary dyskinesia. PLoS One. 2013 Aug 19;8(8):e71409. doi: 10.1371/journal.pone.0071409. eCollection 2013. PMID 23977038
- [Background] Behan L, Rubbo B, Lucas JS, Dunn Galvin A. The patient's experience of primary ciliary dyskinesia: a systematic review. Qual Life Res. 2017 Sep;26(9):2265-2285. doi: 10.1007/s11136-017-1564-y. Epub 2017 Mar 30. PMID 28361274
- [Background] Denizoglu Kulli H, Gurses HN, Zeren M, Ucgun H, Cakir E. Do pulmonary and extrapulmonary features differ among cystic fibrosis, primary ciliary dyskinesia, and healthy children? Pediatr Pulmonol. 2020 Nov;55(11):3067-3073. doi: 10.1002/ppul.25052. Epub 2020 Sep 11. PMID 32877003